CLINICAL TRIAL: NCT02676830
Title: Evaluation of Absorption, Metabolism, and Excretion and Estimation of the Absolute Bioavailability of K-312
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: K-312-1.03US
Record Dates: First submitted 2016-02-02; First posted 2016-02-08 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

ARMS (1):
- K-312 (Experimental)
  Interventions: Drug: K-312 100 mg; Drug: K-312 100 ug C14 IV

INTERVENTIONS:
Drug: K-312 100 mg — Single oral dose
Drug: K-312 100 ug C14 IV — microtracer dose containing ≤37 kBq (1000 nCi) [14C] given as a 5-ml IV push over 2 minutes

SUMMARY:
The purpose of this study is to Evaluation of absorption, metabolism, and excretion of [14C]-K-312 and estimation of the absolute bioavailability of K-312 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study-specific evaluation is performed.
* Subject is a healthy adult male between the ages of 25 and 45 years, inclusive.
* Subject has a body mass index (BMI) of 18.5 to 30 kg/m2, inclusive.

Exclusion Criteria:

* Presence of active or recurring clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease requiring medical treatment.
* Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of K-312.
* Clinically relevant abnormalities in clinical laboratory parameters, as judged by the Investigator.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma-concentration time curve to last measured time point | 336 hours post-dose
Oral bioavailability based on the ratio of AUC after oral dosing to the AUC after i.v. dosing | 336 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Madison, Wisconsin, United States